CLINICAL TRIAL: NCT07301450
Title: An Expanded Access Program of Garetosmab in Patients With Fibrodysplasia Ossificans Progressiva
Brief Title: An Expanded Access Program of Garetosmab in Adult Patients With Fibrodysplasia Ossificans Progressiva (FOP)
Status: Temporarily not available | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R2477-FOP-2081
Record Dates: First submitted 2025-02-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Fibrodysplasia Ossificans Progressiva (FOP)
MeSH Terms: conditions — Myositis Ossificans

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Garetosmab — Administration as described in the protocol
  Other Names: REGN2477

SUMMARY:
The objective of this Expanded Access Program (EAP) is to provide garetosmab to patients with Fibrodysplasia Ossificans Progressiva (FOP) who have completed the double-blind treatment period of the parent study, OPTIMA (R2477-FOP-2175 [NCT05394116]), prior to marketing authorization approval, unless otherwise specified by country specific regulations for rare diseases.

DETAILED DESCRIPTION:
The program will enroll approximately up to 55 patients, globally.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult patients with FOP who must have completed the double-blind treatment period of the parent study OPTIMA (R2477-FOP-2175 [NCT05394116]), as defined in the protocol
2. If the patient has progression of disease with Cumulative Analogue Joint Involvement Scale (CAJIS) >19 at the time of EAP enrollment, the case will require discussion and evaluation between the treating physician and EAP Medical Director to determine final eligibility

Key Exclusion Criteria:

1. Patients participating in OPTIMA who are considered by the treating physician as inappropriate for this program for any reason

NOTE: Other protocol defined inclusion / exclusion criteria apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult